CLINICAL TRIAL: NCT00356525
Title: Phase II, Randomized, Open-Label Trial of Biweekly Pemetrexed Plus Gemcitabine vs. Pemetrexed or Pemetrexed Plus Carboplatin in Relapsed Non Small Cell Lung Cancer After Neoadjuvant or Adjuvant Chemotherapy
Brief Title: Chemotherapy Treatment in Re-occurring Non Small Cell Lung Cancer (NSCLC) After Previous Chemotherapy and Surgical Removal of the NSCLC Tumor
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped early due to low enrollment
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9934; H3E-US-S082 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Results first posted 2009-07-29 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Pemetrexed; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Less Than One Year: Pemetrexed (Experimental): Disease relapse at less than one year after neoadjuvant/adjuvant chemotherapy
  Interventions: Drug: pemetrexed; Drug: gemcitabine
- Less Than One Year: Pemetrexed + Gemcitabine (Experimental): Disease relapse at less than one year after neoadjuvant/adjuvant chemotherapy
  Interventions: Drug: Pemetrexed
- One Year or Greater: Pemetrexed + Carboplatin (Experimental): Disease relapse at one year or greater after neoadjuvant/adjuvant chemotherapy
  Interventions: Drug: carboplatin; Drug: Pemetrexed
- One Year or Greater: Pemetrexed + Gemcitabine (Experimental): Disease relapse at one year or greater after neoadjuvant/adjuvant chemotherapy
  Interventions: Drug: pemetrexed; Drug: gemcitabine

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m2, intravenous (IV), every 14 days x 6 cycles or until disease progression
  Other Names: LY231514; Alimta
  Arms: Less Than One Year: Pemetrexed; One Year or Greater: Pemetrexed + Gemcitabine
Drug: gemcitabine — 1500 mg/m2, intravenous (IV), every 14 days x 6 cycles or until disease progression
  Other Names: LY188011; Gemzar
  Arms: Less Than One Year: Pemetrexed; One Year or Greater: Pemetrexed + Gemcitabine
Drug: carboplatin — area under the curve (AUC) 5, intravenous (IV), every 21 days x 6 cycles or until disease progression
  Arms: One Year or Greater: Pemetrexed + Carboplatin
Drug: Pemetrexed — 500 mg/m2, intravenous (IV), every 21 days x 6 cycles or until disease progression
  Other Names: LY231514; Alimta
  Arms: Less Than One Year: Pemetrexed + Gemcitabine; One Year or Greater: Pemetrexed + Carboplatin

SUMMARY:
The purpose of this study is to help answer:

* Whether pemetrexed, gemcitabine and/or carboplatin can shrink tumor(s) or make tumor(s) disappear in patients with relapsed lung cancer (lung cancer that has come back after surgical removal and chemotherapy), and to determine how long this will last
* Whether pemetrexed, gemcitabine and/or carboplatin can help patients with relapsed lung cancer live longer

ELIGIBILITY:
Inclusion Criteria:

* You have non-small cell lung cancer that has come back (relapsed) after initial treatment with surgery and chemotherapy.
* You have good kidney, liver, and bone marrow organ function.
* You are fully active or able to carry out light work such as housework or office work.

Exclusion Criteria:

* You have received pemetrexed or gemcitabine in the past for lung cancer
* You are currently receiving another treatment for your relapsed lung cancer, or have had chemotherapy or certain other therapies for relapsed lung cancer in the past
* You are unable to take corticosteroid drugs like dexamethasone
* You are unable or unwilling to take the folic acid pills or Vitamin B12 injections that are required for the study
* You are unable to stop taking aspirin or other drugs that control inflammation for certain periods of time during the study
* You have had a heart attack in the last 6 months, or have other heart problems that are not controlled with medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- United States (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evanston, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caxias do Sul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santo André
- India (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trivandrum

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Less Than One Year: Pemetrexed: Disease relapse at less than one year after neoadjuvant/adjuvant chemotherapy. Pemetrexed: 500 mg/m2, intravenous (IV), every 21 days x 6 cycles or until disease progression
- Less Than One Year: Pemetrexed + Gemcitabine: Disease relapse at less than one year after neoadjuvant/adjuvant chemotherapy. Pemetrexed: 500 mg/m2, intravenous (IV), every 14 days x 6 cycles or until disease progression Gemcitabine: 1500 mg/m2, IV, every 14 days x 6 cycles or until disease progression
- One Year or Greater: Pemetrexed + Carboplatin: Disease relapse at one year or greater after neoadjuvant/adjuvant chemotherapy. Pemetrexed: 500 mg/m2, intravenous (IV), every 21 days x 6 cycles or until disease progression Carboplatin: Area under the curve (AUC) 5, intravenous (IV), every 21 days x 6 cycles or until disease progression
- One Year or Greater: Pemetrexed + Gemcitabine: Disease relapse at one year or greater after neoadjuvant/adjuvant chemotherapy. Pemetrexed: 500 mg/m2, intravenous (IV), every 14 days x 6 cycles or until disease progression Gemcitabine: 1500 mg/m2, IV, every 14 days x 6 cycles or until disease progression
Period: Overall Study
Arm/Group | Less Than One Year: Pemetrexed | Less Than One Year: Pemetrexed + Gemcitabine | One Year or Greater: Pemetrexed + Carboplatin | One Year or Greater: Pemetrexed + Gemcitabine
Started | 14 | 11 | 7 | 9
Completed | 0 | 0 | 0 | 0
Not Completed | 14 | 11 | 7 | 9
Not completed — Progressive Disease | 8 | 5 | 4 | 2
Not completed — Adverse Event | 1 | 3 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 2 | 2 | 1
Not completed — Protocol Entry Criteria Not Met | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 3
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Sponsor Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Less Than One Year: Pemetrexed | Less Than One Year: Pemetrexed + Gemcitabine | One Year or Greater: Pemetrexed + Carboplatin | One Year or Greater: Pemetrexed + Gemcitabine | Total
Number analyzed (Participants) | 14 | 11 | 7 | 9 | 41
Age, Customized [Number; unit: participants]
  <=65 years | 6 | 3 | 2 | 4 | 15
  >65 years | 8 | 8 | 5 | 5 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 0 | 4 | 16
  Male | 8 | 5 | 7 | 5 | 25
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 7 | 9 | 41
Disease Stage at Initial Diagnosis [Number; unit: participants] — Stages of disease range from 0 (no evidence of primary tumor) to IV (tumor in multiple locations).
  participants
    Stage IV | 14 | 11 | 7 | 9 | 41
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 6 | 3 | 2 | 6 | 17
    1 - Ambulatory, Restricted Strenuous Activity | 8 | 8 | 5 | 3 | 24
History of Brain Metastates [Number; unit: participants]
  No | 12 | 11 | 7 | 9 | 39
  Yes | 2 | 0 | 0 | 0 | 2
Prior Systemic Therapy [Number; unit: participants] — Participants could have more than one type of prior systemic therapy which may result in the total numbers per arm being larger than the overall number of participants per arm.
  participants
    Adjuvant | 12 | 11 | 6 | 9 | 38
    Neoadjuvant | 3 | 0 | 1 | 1 | 5
Race/Ethnicity [Number; unit: participants]
  Black or African American | 0 | 0 | 2 | 0 | 2
  East Asian | 0 | 0 | 0 | 1 | 1
  West Asian | 0 | 0 | 0 | 1 | 1
  Caucasian | 14 | 11 | 5 | 7 | 37

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response
Description: Best response recorded from the start of treatment until disease progression/recurrence using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria.
Time Frame: baseline to time of response (up to 17.5 months)
Population: Number of randomized participants in each category.
Measure: Number; unit: participants
Arm/Group | Less Than One Year: Pemetrexed | Less Than One Year: Pemetrexed + Gemcitabine | One Year or Greater: Pemetrexed + Carboplatin | One Year or Greater: Pemetrexed + Gemcitabine
Number analyzed (Participants) | 14 | 11 | 7 | 9
participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 7 | 0 | 2 | 1
  Stable Disease | 3 | 9 | 5 | 6
  Progressive Disease | 2 | 2 | 0 | 1
  Unknown | 2 | 0 | 0 | 1

2. Secondary Outcome: Overall Survival
Description: Overall survival is the number of participants who were alive when the trial was terminated.
Time Frame: baseline to trial termination (17.5 months)
Population: Number of randomized participants in each category.
Measure: Number; unit: participants alive
Arm/Group | Less Than One Year: Pemetrexed | Less Than One Year: Pemetrexed + Gemcitabine | One Year or Greater: Pemetrexed + Carboplatin | One Year or Greater: Pemetrexed + Gemcitabine
Number analyzed (Participants) | 14 | 11 | 7 | 9
participants alive | 6 [1.64 to 16.10] | 4 [0.99 to 11.66] | 6 [4.40 to 17.58] | 7 [0.16 to 14.78]

3. Secondary Outcome: Time to Progressive Disease
Time Frame: baseline to measured progressive disease (up to 17.5 months)
Population: Outcome measure was not analyzed due to insufficient data.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Less Than One Year: Pemetrexed | Less Than One Year: Pemetrexed + Gemcitabine | One Year or Greater: Pemetrexed + Carboplatin | One Year or Greater: Pemetrexed + Gemcitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Duration of Response
Time Frame: time of response to progressive disease (up to 17.5 months)
Population: Outcome measure was not analyzed due to insufficient data.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Less Than One Year: Pemetrexed | Less Than One Year: Pemetrexed + Gemcitabine | One Year or Greater: Pemetrexed + Carboplatin | One Year or Greater: Pemetrexed + Gemcitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Time to Treatment Failure
Time Frame: baseline to stopping treatment (up to 17.5 months)
Population: Outcome measure was not analyzed due to insufficient data.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Less Than One Year: Pemetrexed | Less Than One Year: Pemetrexed + Gemcitabine | One Year or Greater: Pemetrexed + Carboplatin | One Year or Greater: Pemetrexed + Gemcitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Less Than One Year: Pemetrexed | Less Than One Year: Pemetrexed + Gemcitabine | One Year or Greater: Pemetrexed + Carboplatin | One Year or Greater: Pemetrexed + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 3/14 | 5/11 | 0/7 | 2/9
Other Adverse Events (participants affected / at risk) | 14/14 | 11/11 | 7/7 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Less Than One Year: Pemetrexed (N=14) | Less Than One Year: Pemetrexed + Gemcitabine (N=11) | One Year or Greater: Pemetrexed + Carboplatin (N=7) | One Year or Greater: Pemetrexed + Gemcitabine (N=9)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Less Than One Year: Pemetrexed (N=14) | Less Than One Year: Pemetrexed + Gemcitabine (N=11) | One Year or Greater: Pemetrexed + Carboplatin (N=7) | One Year or Greater: Pemetrexed + Gemcitabine (N=9)
Anaemia (Blood and lymphatic system disorders) | 6 (10) | 10 (15) | 1 (3) | 3 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (4) | 0 (0) | 1 (3)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 4 (4) | 2 (8) | 3 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 4 (4) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Porokeratosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye allergy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (7) | 6 (6) | 3 (4) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (8) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (15) | 6 (10) | 3 (7) | 6 (10)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 4 (4) | 1 (2) | 3 (4)
Asthenia (General disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 11 (17) | 11 (21) | 5 (7) | 6 (6)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal dryness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (5) | 5 (7) | 0 (0) | 2 (3)
Secretion discharge (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Collapse of lung (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 1 (2)
Aspiration pleural cavity (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (5)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prothrombin time ratio (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sputum culture positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (4)
White blood cell count increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 2 (3) | 2 (4) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 4 (7) | 2 (2) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (3) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 1 (1) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 5 (6) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Radial nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 4 (9) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 6 (9) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4) | 2 (2) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 4 (6) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (7) | 4 (5) | 3 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (7) | 2 (3) | 2 (2)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mechanical ventilation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thoracotomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 6 (6) | 5 (5) | 5 (5)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial terminated early due to slow enrollment. Secondary outcomes were not analyzed due to insufficient data. Original results reported were interim analyses. Results have now been updated with final data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days